CLINICAL TRIAL: NCT02889731
Title: The "Suicide Guard Rail": A Structural Intervention for Hospitals Avoid Suicides by Jumping From Heights Buildings
Status: Completed | Type: Observational
Sponsor: Kantonsspital Baden (Other)
Collaborators: Police department at Baden (Unknown)
Responsible Party: Principal Investigator, Juerg H. Beer, Prof. Dr. med, Kantonsspital Baden
Other Study IDs: IRB 11/06
Record Dates: First submitted 2015-09-21; First posted 2016-09-07 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-08

CONDITIONS: Suicide Jumps; Psychiatry
Keywords: Suicide; Heights; Suicide hot spots; Bridges
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background: Suicides by jumping from the high buildings of acute hospitals are dramatic events which are highly traumatizing to families, staff and fellow pts. In the 10 years from1995 to 2010 the investigators have counted 10 suicide cases despite extensive measures taken to predict and avoid them.

The investigators hypothesized that constructive measures at the windows that would render access more difficult could discourage spontaneous suicidal behaviour and would reduce the suicide rates.

Intervention: Starting in 6/2004, a 20 mm diameter metal guard-rail (which resists 250kg) was installed at each window of a 360 bed acute hospital at a height of 113cm, 18cm above the window parapet with the aim to visually, psychologically and physically discourage potential suicidal impulses.

ELIGIBILITY:
Inclusion Criteria:

* person at risk for suicide

Exclusion Criteria:

* no

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: in-patients and out-patients
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2004-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Number of Suicide Jumps over ten years | Between 1995 and 2010, measurement 180 months
  Suicide jumps from the heights of acute hospitals are dramatic events which are highly traumatizing to families, staff, and fellow patients. From 1995 to 2004, 10 suicide jumps occurred at the investigators institution despite extensive measures taken to predict and avoid them. The investigators hypothesized that specific barriers rendering access to windows more difficult could discourage spontaneous suicidal behaviour and reduce the suicide rates. Starting in 6/2004, a 20 mm diameter metal guard-rail with a tension strength of 250kg/in2 was installed at each window of the investigators 360 bed acute hospital at a height of 113cm, 18cm above the window sill with the aim to psychologically and physically deter potential suicidal impulses.